CLINICAL TRIAL: NCT00293605
Title: Effect of Cemented Stem Design on Periprosthetic Bone Mass Following Primary Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Mr Andrew Hamer, Sheffield NHS Foundation Trust
Other Study IDs: NS200361715
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Osteoarthritis
Keywords: aseptic loosening; femoral stem design
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: C-stem implant
  Interventions: Procedure: Total Hip Replacement
- 2: Charnley Implant
  Interventions: Procedure: Total Hip Replacement
- 3: Exeter Implant
  Interventions: Procedure: Total Hip Replacement

INTERVENTIONS:
Procedure: Total Hip Replacement — Implantation of one of 3 stem designs

SUMMARY:
Total hip replacement is a common procedure for the treatment of osteoarthrosis of the hips, the aims of this study are to determine the effect of implant stem design on bone quality surrounding the implant using three stem designs that are routinely implanted at this hospital.

DETAILED DESCRIPTION:
120 patients will undergo routine hip replacements using either the C-Stem, Exeter Stem or Charnley stem implants. Patients will be clinically evaluated pre-operatively and randomised to one of the three implants. Post-operatively, patients will be clinically reviewed for 2 years using bone mineral density scans, radiological review, blood and urine analysis for bone markers and validated questionnaires to assess clinical data (Oxford Hip and Harries Hip). Patients will be assessed for prothesis migration using the EBRA methods.

ELIGIBILITY:
Inclusion Criteria:

* patients must be aged 60 yrs or more uncomplicated primary or secondary osteoarthritis of the hip undergoing unilateral cemented total hip arthroplasty using a metal on polyethylene bearing couple.

Exclusion Criteria:

* metabolic bone disorders, systemic disorders such as rheumatoid arthritis and patients who have taken pharmacological doses of oral steroids, hormone replacement therapy, tamoxifen, calcium or vitamin D supplements within the last year. Patients with a prior history of bisphosphonates and women of child bearing age.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-assessment clinics at Sheffield Hospitals, patients booked for hip replacements.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2004-01; Primary Completion 2008-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Proximal femoral BMD change over 2 years measured by DXA | 2 years

SECONDARY OUTCOMES:
Clinical Evaluation using patient centered questionnaire (Oxford Hip Score) | 2 years
Surgeon centered clinical assessment (Harris Hip Score) | 2 years
Plain radiographic assessment | 2 years
Biochemical markers of bone formation and resorption measured from serum and urine samples using the Elecsys system. | 2 years
Femoral prosthetic stem y-axis migration (subsidence), ans stem/shaft angulation change measured by EBRA. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Hamer, FRCS, Principal Investigator — STH NHS Foundation Trust
Locations (1):
- Orthopaedic Department, Northern General Hospital, Sheffield, South Yorkshire, United Kingdom